CLINICAL TRIAL: NCT03951493
Title: Phase III Randomized, Controlled, Open, Multicentre Medical-economic Study Evaluating the Efficacy of Adding ZOlédronique Acid to STERéotaxique Radiotherapy in the Treatment of Vertebral Metastases
Brief Title: Multicentre Medical-economic Study Evaluating the Efficacy of Adding ZOlédronique Acid to STERéotaxique Radiotherapy in the Treatment of Vertebral Metastases
Acronym: ZOSTER
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICO-N-2018-14
Record Dates: First submitted 2019-05-10; First posted 2019-05-15 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Vertebral Metastasis
Keywords: Hypo-fractured radiotherapy in stereotactic conditions (RSHF); zoledronic acid; medico-economic; vertebral compressive fracture
MeSH Terms: interventions — Zoledronic Acid; Solutions; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RSHF + zoledronic acid (Experimental): Patients receive RSHF according to : 30 Gy in 5 fractions of 6 Gy spaced 48 hours or 27 Gy in 3 fractions of 9 Gy spaced 48 hours or 20 Gy in 1 fraction. combined with zoledronic acid (4 mg IV slow monthly for 12 months, dose adjusted according to creatinine clearance).
  Interventions: Combination Product: Zoledronic Acid 4Mg Solution for Injection + Hypo-fractured radiotherapy in stereotactic conditions
- RSHF (Active Comparator): Patients receive only RSHF according to : 30 Gy in 5 fractions of 6 Gy spaced 48 hours or 27 Gy in 3 fractions of 9 Gy spaced 48 hours or 20 Gy in 1 fraction.
  Interventions: Radiation: Hypo-fractured radiotherapy in stereotactic conditions

INTERVENTIONS:
Combination Product: Zoledronic Acid 4Mg Solution for Injection + Hypo-fractured radiotherapy in stereotactic conditions — All patients receive radiotherapy i.e. treatment on D1, D3 and D5.
  Several radiotherapy schemes are possible:
  * 20 Gy in 1 fraction;
  * 27 Gy in 3 fractions of 9 Gy
  * 30 Gy in 5 fractions of 6 Gy. All patients in the experimental arm receive an intravenous injection of at least 15 minutes of 4 mg zoledronic acid every month for 12 months.
  The first injection must be made no more than 3 weeks before the first day of radiotherapy. It can be performed up to J1 of radiotherapy.
  The injections will be carried out either at the patient's home by the nurses or in the investigator centre.
  Arms: RSHF + zoledronic acid
Radiation: Hypo-fractured radiotherapy in stereotactic conditions — All patients receive radiotherapy i.e. treatment on D1, D3 and D5.
  Several radiotherapy schemes are possible:
  * 20 Gy in 1 fraction;
  * 27 Gy in 3 fractions of 9 Gy
  * 30 Gy in 5 fractions of 6 Gy.
  Arms: RSHF

SUMMARY:
Hypo-fractured radiotherapy in stereotactic conditions (RSHF) of bone metastases allows high doses to be delivered to the affected bone segment while sparing adjacent healthy tissues as well as possible. In addition, it not only reduces pain and prevents spinal cord compression, but also improves long-term control of metastatic disease.

Zoledronic acid reduces bone complications. The economic literature shows that stereotactic radiotherapy, like zoledronic acid, are cost-effective strategies in these indications. The objective of this research project is to evaluate the efficiency of adding zoledronic acid to stereotactic radiotherapy in the treatment of vertebral metastases.

ELIGIBILITY:
Inclusion Criteria:

* Cancer with inoperable thoracic and/or lumbar vertebral metastasis;
* Age ≥ 18 years old ;
* Life expectancy greater than 1 year;
* OMS or PS ≤ 2 ;
* Effective contraception for women of childbearing age;
* Patient information and free, informed and written consent, signed by the patient and investigator;
* Patient affiliated or beneficiary of the social security system.

Exclusion Criteria:

* Cancer with inoperable thoracic and/or lumbar vertebral metastasis;
* Painful patient unable to maintain a lying position for 30 minutes despite analgesic treatment;
* Patient who has received external irradiation from the proposed irradiation area > 20 Gy ;
* Signs of neurological compression;
* Spinal cord compression or epidural damage requiring surgery before radiotherapy;
* Clinically significant hypersensitivity to zoledronic acid, other bisphosphonates or any excipient;
* History of osteonecrosis of the maxilla or bone exposure or delayed healing after dental surgery;
* Previous (less than 2 years) or ongoing treatment with a bisphosphonate;
* Creatinine clearance < 30 ml/min;
* Pregnant or breastfeeding woman;
* Patient protected or under guardianship or incapable of giving consent;
* Impossibility to submit to the medical follow-up of the trial for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2020-06-23 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Differential Cost Result Ratio (DCRR) expressed as cost per year of life earned in good health | 24 months
  The determination of the DCRR includes Identification of care consumption ; The measurement of costs ; overall survival at 2 years ; Calculation of utilities using the EQ5D-5L questionnaire

SECONDARY OUTCOMES:
Survival without vertebral compression fractures | At 12 months and 24 months
Pain control | at inclusion, 12 and 24 months
  Pain control will be assessed using a visual analogue scale (VAS) that measures pain intensity, prevents it, initiates or monitors drug or non-drug treatment, and the Brief Pain inventory, a questionnaire that quickly assesses the severity of pain and its impact on the patient's daily life.
Survival without bone complication | At 12 months and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane SUPIOT, MD, Study Director — ICO site SAINT HERBLAIN
Locations (7):
- France (7):
  - Institut BERGONIE, Bordeaux
  - Institut de Cancérologie de Lorraine, Nancy
  - Hôpital Privé du Confluent, Nantes
  - Centre de Haute Energie, Nice
  - Hopital Lyon Sud, Pierre-Bénite
  - Centre Henri Becquerel, Rouen
  - Stéphane SUPIOT, Saint-Herblain